CLINICAL TRIAL: NCT00432536
Title: Redesigning Cardiac Surgery to Reduce Neurologic Injury
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: MaineHealth (Other); Catholic Medical Center (Other); Somanetics Corporation (Industry); LivaNova (Industry); Maquet Cardiovascular (Industry); Northern New England Cardiovascular Disease Study Group (Unknown); Luna Innovations (Industry); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David J. Malenka, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: 20307; 1K02HS015663-01A1 (AHRQ)
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Disease; Surgery
Keywords: Neuro-monitoring; Quality Improvement; Cerebral emboli; Cerebral desaturation; Hypotension
MeSH Terms: conditions — Cardiovascular Diseases; Intracranial Embolism; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum to study neurologic biomarker, Sb100.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quality improvement intervention — determine the effectiveness of adopting quality improvement strategies to reduce embolization, hypotension and cerebral desaturation

SUMMARY:
Neurologic injuries are frequent and devastating complications following cardiac surgery. Previous work conducted by our research group and others has identified the principal mechanisms creating both overt and subtle neurologic injuries after cardiac surgery. Current work by our group has identified that the causes (thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli) of these injuries are byproducts of processes of surgical and perfusion care. This insight suggests that the redesign of clinical strategies and techniques to prevent the occurrence of these intraoperative sources of damage may provide an opportunity to reduce the risk of neurologic injury after cardiac surgery.

The goal of this research is to identify modifiable clinical strategies and techniques of surgical and perfusion care associated with the causes (thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli) of neurologic injury secondary to coronary artery bypass graft (CABG) surgery, and subsequently to redesign these processes to reduce a patient's risk of a neurologic injury.

DETAILED DESCRIPTION:
The goal of this research is to identify modifiable clinical strategies and techniques of surgical and perfusion care associated with the causes (thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli) of neurologic injury secondary to coronary artery bypass graft (CABG) surgery, and subsequently to redesign these processes to reduce a patient's risk of a neurologic injury. The following hypotheses will be addressed.

Hypothesis #1a. Identifying alternative strategies for conducting processes of surgical and perfusion care will reveal opportunities to reduce the occurrence of causes of neurologic injury. The most common mechanisms creating neurologic injury, whether focal or global, after CABG surgery are thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli. Processes of surgical and perfusion care are associated with the creation of each of these causes of neurologic injury.

Hypothesis #1b. Redesigning processes of surgical and perfusion care to reduce thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli during CABG surgery will result in reductions of tissue-level and neurologic injury. We will analyze sera for tissue-level brain injury as well as identify any new neurologic injuries present among patients undergoing CABG surgery. Redesigning CABG surgery to reduce thrombotic/lipid emboli, cerebral hypoperfusion & hypotension, and gaseous emboli will result in decreases in tissue-level and neurologic injury.

Hypothesis #2. A regional quality improvement intervention will result in changes to surgical and perfusion techniques. Regional dissemination of the findings from Hypotheses #1a,b may be realized through focused quality improvement initiatives utilizing multidisciplinary clinical teams.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-89 years undergoing nonemergency coronary revascularization or valve procedures with or without the use of a cardiopulmonary bypass circuit.

Exclusion Criteria:

- Undergoing concomitant procedures besides cardiac surgery

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2002-10; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Emboli and Hypoperfusion Counts | within the operative time period
  We will count the number of thrombotic/lipid emboli and number of gaseous emboli. Along with the number of hypotensive events. We will link counts to surgical and perfusion techniques.

SECONDARY OUTCOMES:
Type I and II neurologic injuries | within 3 months after surgery
  We will measure a patient's neurologic status Using a Telephone Interview for Cognitive Status tool at 3 time periods (prior to surgery, prior to discharge and at 3 months)
Tissue-level neurologic injury | within 48 hrs of surgery
  Blood for serum markers will be collected after surgery. We will assess plasma levels of biochemical markers of neurology injury.

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Likosky, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; David J. Malenka, MD, Study Director — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Maine Medical Center, Portland, Maine
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire

REFERENCES:
- [Result] Likosky DS, Donegan DJ, Groom RC, Buchanan SA, Morton JR, Ross CS, O'Connor GT. Embolic activity subsequent to injection of the internal mammary artery with papaverine hydrochloride. Heart Surg Forum. 2005;8(6):E434-6. doi: 10.1532/HSF98.20051012. PMID 16283980
- [Result] Likosky DS, Groom RC, Clark C, Forest RJ, Kramer RS, Morton JR, Ross CS, Sabadosa KA, O'Connor GT; Northern New England Cardiovascular Disease Study Group, Lebanon, New Hampshire. A method for identifying mechanisms of neurologic injury from cardiac surgery. Heart Surg Forum. 2004;7(6):348-52. doi: 10.1532/HSF98.20041088. PMID 15769702
- [Result] Groom R, Likosky DS, Rutberg H. Understanding variation in cardiopulmonary bypass: Statistical Process Control Theory. J Extra Corpor Technol. 2004 Sep;36(3):224-30. No abstract available. PMID 15559738
- [Result] Groom RC, Likosky DS, Forest RJ, O'Connor GT, Morton JR, Ross CS, Clark C, Kramer R. A model for cardiopulmonary bypass redesign. Perfusion. 2004 Jul;19(4):257-61. doi: 10.1191/0269216304pf749oa. PMID 15376771
- [Result] Groom RC, Quinn RD, Lennon P, Welch J, Kramer RS, Ross CS, Beaulieu PA, Brown JR, Malenka DJ, O'Connor GT, Likosky DS; Northern New England Cardiovascular Disease Study Group. Microemboli from cardiopulmonary bypass are associated with a serum marker of brain injury. J Extra Corpor Technol. 2010 Mar;42(1):40-4. PMID 20437790
- [Result] Groom RC, Quinn RD, Lennon P, Donegan DJ, Braxton JH, Kramer RS, Weldner PW, Russo L, Blank SD, Christie AA, Taenzer AH, Forest RJ, Clark C, Welch J, Ross CS, O'Connor GT, Likosky DS; Northern New England Cardiovascular Disease Study Group. Detection and elimination of microemboli related to cardiopulmonary bypass. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):191-8. doi: 10.1161/CIRCOUTCOMES.108.803163. Epub 2009 May 5. PMID 20031837